CLINICAL TRIAL: NCT02012595
Title: [11C]Donepezil PET For Imaging The Autonomous Nervous System In Parkinsons Disease
Status: Completed | Type: Observational
Sponsor: Per Borghammer (Other)
Collaborators: Lundbeck Foundation (Other); Jascha Fonden (Other); Fonden af 2. Juli 1984 til bekæmpelse af Parkinsons Sygdom, Denmark (Other)
Responsible Party: Sponsor-Investigator, Per Borghammer, MD, ph.d.,DMSci, Aarhus University Hospital
Organization: University of Aarhus (Other)
Other Study IDs: 2013-01; 2013-003775-35 (EudraCT Number)
Record Dates: First submitted 2013-11-26; First posted 2013-12-16 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2015-05

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Parkinson's patients: Participants with Parkinson's Disease
  Interventions: Other: [11C]donepezil PET
- Healthy Controls: Healthy participants
  Interventions: Other: [11C]donepezil PET

INTERVENTIONS:
Other: [11C]donepezil PET — Positon Emission Tomography (PET) imaging of acetylcholinesterase using the ligand [11C]donepezil

SUMMARY:
AIM: Investigate wether there are differences in the parasympathetic nervous system in Parkinsons patients compared to controls.

MATERIALS AND METHODS: We use the tracer [11C]donepezil to image the parasympathetic nervous system. The Investigators will include 20 Parkinsons patients and 20 healthy controls aged 40-80 in our study. The participants will receive a careful medical examination, including a neurological examination, as part of the inclusion process. The subjects also have an MRI scan of the brain. Then PET/CT scans with [11C]donepezil are conducted - once for the upper abdominal region and once for the head region. For evaluating the function of the parasympathetic nervous system gastric emptying time, heart rate variability and salivary flow will be measured. These measureless will be correlated to the PET findings.

PERSPECTIVES: The study will potentially result in the development of a PET ligand for imaging the parasympathetic nervous system. This will have applications for research in Parkinson's disease, diabetes, heart disease and other disorders, in which the autonomic nervous system is involved

ELIGIBILITY:
Inclusion Criteria:

* Age 40-80 years

Exclusion Criteria:

* dementia,
* psychiatric diseases,
* serious medical illness including any type of previous cancer
* any drug with known interaction with the autonomic nervous system
* metal in the body (because of MRI scan)
* pregnancy or breast feeding (because of radiation due to PET/CT)
* known diseases of the salivary glands, stomach, intestines.
* Prior major surgery to salivary glands, esophagus, stomach.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Parkinson's patients with moderate symptoms (diagnosis > 4 years earlier, bilateral disease). Will be recruited through department of neurology Aarhus University Hospital, Denmark.
  Healthy controls recruited through local media.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2013-10; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Distribution volume of [11C]donepezil in internal organs | The distribution volume of [11C]donepezil is measured at "Day 1" by PET/CT scanning each participant. The data analysis is done when all participants have completed the study.
  Our primary endpoint is the distribution volume of [11C]donepezil in internal organs (including salivary glands, heart, stomach and intestines) in Parkinson's patients compared to controls.

CONTACTS AND LOCATIONS:
Overall Officials: Per Borghammer, MD, PhD,DMSc, Principal Investigator — Dept. of Nuclear Medicine & PET Center, Aarhus University Hospital, Aarhus, Denmark
Locations (1):
- Dept. of Nuclear Medicine & PET Center, Aarhus University Hospital, Aarhus, Denmark